CLINICAL TRIAL: NCT01893125
Title: A Randomised Three Week Double-blind Crossover Study to Compare the Efficacy and Safety of CNV2197944 75 mg Tid Versus Placebo in the Treatment of Neuropathic Pain in Patients With Diabetic Peripheral Neuropathy
Brief Title: Efficacy and Safety of CNV2197944 Versus Placebo in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Convergence Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CNV2197944/202
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNV2197944 (Experimental): CNV2197944 75mg tid 21 days
  Interventions: Drug: CNV2197944
- Placebo (Placebo Comparator): Placebo 1 cap tid 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNV2197944
  Arms: CNV2197944
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate the effect of repeat oral dosing of CNV2197944 75 mg tid on the pain experienced in diabetic peripheral neuropathy (DPN) as measured by changes in PI-NRS after three weeks of treatment compared to the baseline period.

DETAILED DESCRIPTION:
A 3 week randomised crossover study to investigate the effect of repeat oral dosing of CNV2197944 75 mg tid versus placebo for on the pain experienced in diabetic peripheral neuropathy (DPN). Each 3 week treatment period is seperated by a 2 week washout period. The primary outcome measure is the change from baseline in the PI-NRS after three weeks of treatment. Secondary outcome measures include pain responder rates, clinical and patient global impressions of pain, and the Neuropathic Pain Symptom Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 85 years of age inclusive, at the time of signing the informed consent
* Diabetes Mellitus (Type I or II)with HbA1c <9%
* Evidence of symmetrical bilateral pain in lower limbs with evidence of decreased sensation or impaired reflexes and a Michigan Neuropathy Screening -Instrument score of >3 on physical examination
* Patients with diabetic peripheral neuropathy (DPN) with pain at screening present for more than 6 months. The maximum duration of DPN will be no longer than 5 years

Exclusion Criteria:

* Patients having other severe pain, which may impair the self-assessment of the pain due to DPN
* Patients who have received nerve blocks for neuropathic pain within 4 weeks -Patients on other concomitant medications used to relieve the pain of DPN
* Patients with a documented failure to respond to a maximally tolerated dose regimen of gabapentin or pregabalin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Numerical Rating Scale | 21 days

SECONDARY OUTCOMES:
Pain Responder rates | 21 days
Neuropathic Pain Symptom Inventory | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Hidvegi, MD, PhD, Principal Investigator — Dept. Metabolism and Diabetes, Gyor, Hungary
Locations (1):
- Petz Aladar County Teaching Hospital, Győr, Gyor, Hungary